CLINICAL TRIAL: NCT01361620
Title: Genotypic and Phenotypic Correlates of Resistance to Anti-platelet Actions of Aspirin in an At-risk Patient Population and in the General Population
Brief Title: Genotypic and Phenotypic Correlates of Resistance to Aspirin
Acronym: ARSENAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: George Washington University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: AR2011
Record Dates: First submitted 2011-05-25; First posted 2011-05-27 (Estimated); Results first posted 2013-12-16 (Estimated); Last update posted 2013-12-16 (Estimated); Status verified 2011-01

CONDITIONS: Platelet Dysfunction Due to Aspirin
Keywords: genomic markers; aspirin resistance
MeSH Terms: interventions — Aspirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Aspirin (Other): All subjects took 7-10 days of 81 mg aspirin
  Interventions: Drug: aspirin

INTERVENTIONS:
Drug: aspirin — aspirin 81mg, 7-10 days

SUMMARY:
The study seeks to identify genomic markers associated with aspirin resistance.

DETAILED DESCRIPTION:
Not desired

ELIGIBILITY:
Inclusion Criteria:

* Volunteers 40 to 80 years old willing to sign consent and take 81 mg of aspirin for 7 - 10 days and return for laboratory testing.

Exclusion Criteria:

* Patient requiring more than 81 mg aspirin daily
* Known GI bleeding attributed to ASA
* Active peptic ulcer disease or history within the last year
* Known aspirin allergy
* Current use of:

  * warfarin,
  * heparin,
  * NSAIDs (except aspirin),
  * clopidogrel,
  * dipyridamole,
  * fish-oil/omega 3 supplements,
* Women of childbearing potential who are pregnant, planning to become pregnant or nursing.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 190 (Actual)
Dates: Start 2007-12; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Reiner, MD, Principal Investigator — GWU Medical Faculty
Locations (1):
- GWU Medical Faculty Associates, Washington D.C., District of Columbia, United States

REFERENCES:
- [Result] Fallahi P, Katz R, Toma I, Li R, Reiner J, VanHouten K, Carpio L, Marshall L, Lian Y, Bupp S, Fu SW, Rickles F, Leitenberg D, Lai Y, Weksler BB, Rebling F, Yang Z, McCaffrey TA. Aspirin insensitive thrombophilia: transcript profiling of blood identifies platelet abnormalities and HLA restriction. Gene. 2013 May 15;520(2):131-8. doi: 10.1016/j.gene.2013.02.032. Epub 2013 Feb 27. PMID 23454623

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from patients of the GWU Medical Faculty Associates, and physicians, faculty and staff on the GWU campus. Initially we were looking for those already prescribed to take aspirin at 81 mg daily, but due to slow recruitment, this was amended to anyone willing to take aspirin at 81 mg daily for 7-10 days
Pre-assignment Details: Excluded were 58 subjects prescribed more than 81 mg of aspirin, had known GI bleeding attributed to aspirin, active peptic ulcer disease, aspirin allergy, current use of other anti-platelet, anti-thrombotic or other therapy that has these properties, women who are pregnant, planning pregnancy or nursing. Exclusions were for safety reasons.
Period: Overall Study
Arm/Group | Aspirin
Started | 132
Completed | 132
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Aspirin
Number analyzed (Participants) | 132
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 91
  >=65 years | 41
Age Continuous [Mean (Standard Deviation); unit: years] | 61 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52
  Male | 80
Region of Enrollment [Number; unit: participants]
  United States | 132

OUTCOME MEASURES:

1. Primary Outcome: Whole Blood Coagulation
Description: Whole blood coagulation after stimulation with arachidonic acid, as measured in the VerifyNow Aspirin system (Accumetrics). Aspirin response units (ARU) are the residual coagulation present in patients taking aspirin. The higher the ARU, the greater residual coagulation (resistance) to the aspirin effect.
Time Frame: Single measurement at 7-10 days after beginning aspirin
Measure: Mean (Standard Deviation); unit: Aspirin response units (ARU)
Arm/Group | Aspirin
Number analyzed (Participants) | 132
Aspirin response units (ARU) | 453.8 (51.9)

ADVERSE EVENTS:
Arm/Group | Aspirin
Serious Adverse Events (participants affected / at risk) | 0/132
Other Adverse Events (participants affected / at risk) | 0/132

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No